CLINICAL TRIAL: NCT00753610
Title: Effect of Concurrent Chemoradiation on Circulating Endothelial Progenitor Cells in Cervical Cancer
Brief Title: Endothelial Progenitor Cells in Cervical Cancer Patients Receiving Chemoradiation
Acronym: EPC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Yu-Jen Chen, Head, Department of Radiation Oncology, Mackay Memorial Hospital
Other Study IDs: MMH-I-S-354
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Cervical Cancer
Keywords: EPC; CCRT; Cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Invasive carcinoma of the uterine cervix remains the most common invasive cancer in women in many countries. Concurrent chemoradiotherapy (CCRT) is now recommended as a standard treatment for locally advanced and high-risk cervical carcinoma. However, CCRT achieves a better control of cervical cancer accompanied by greater morbidity. To avoid unnecessary over-treatment, the optimization of CCRT is of critical importance. Herein, the development of a surrogate marker for monitoring treatment efficacy as well as toxicity is pivotal to optimize CCRT.

Circulating endothelial progenitor cells (EPC), derived from bone marrow, can be used as a marker for optimizing and monitoring the anti-angiogenesis therapy including angiogenesis inhibitors and metronomic chemotherapy. Preclinical models indicated that the source of apoptotic circulating endothelial cells (CEC) was most likely the tumor vasculature. In breast cancer patients, apoptotic CEC were demonstrated to be a surrogate marker for efficacy of metronomic therapy.

In this grant, we intent to monitor the levels of circulating EPC/CEC in locally advanced cervical cancer patients before, during and after CCRT.

DETAILED DESCRIPTION:
Invasive carcinoma of the uterine cervix remains the most common invasive cancer in women in many countries. Concurrent chemoradiotherapy (CCRT) is now recommended as a standard treatment for locally advanced and high-risk cervical carcinoma (1-3). Although the local control rate and survival have improved with use of CCRT, the treatment does cause greater toxicity in the bone marrow and other normal tissues compared with that caused by conventional RT. Our previous study demonstrated that serial changes in serum cytokines during chemoradiation correlated with tumor regression and treatment morbidity. The sudden elevation of serum TGF-beta 1 and VEGF levels after the first fraction of brachytherapy correlate with the development of greater RT morbidity. Higher pretreatment TGF-beta 1 and VEGF levels are associated with poor tumor response to chemoradiation (4). It implicates that angiogenic factor, such as VEGF, may play roles in the toxicity and outcome of CCRT. However, it still lacks a surrogate marker for prediction of clinical outcome of CCRT.

The most commonly used chemotherapeutic drugs combined with radiation as radiosensitizers are cis-platinum and 5-fluorouracil. These drugs, especially cis-platinum, are toxic to kidney, myelosuppressive and prone to cause life-threatening neutropenia, anemia or thrombocytopenia, which are more severe than those with radiotherapy alone (1-3). To avoid unnecessary over-treatment, the optimization of CCRT is of critical importance. Herein, the development of a surrogate marker for monitoring treatment efficacy as well as toxicity is pivotal to optimize CCRT.

Angiogenesis is a heavily regulated process, which is involved by complex interactions between inhibitory and stimulatory angiogenic factors. It is essential for tumor growth, progression and metastasis and is correlated with poor prognosis in cancer patients including cervical cancer (5). Many novel compounds, such as EGCG (6), that potently inhibit formation of neoplastic blood vessels have been recently developed. There is increasing interest in developing angiogeneis-suppressive agents for cancer treatment and growing number of anti-angiogenesis drugs currently being evaluated in clinical trials for various malignancies. Promising results have been reported include an increase in overall survival and reduction in the risk of death (Bevacizumab), reversal of cellular drug resistance (Cetuximab) and activity as second-line therapy in colorectal cancer patients who have exhausted other available treatment options (Cetuximab, ABX-EGF, PTK-787, Gefitinib, Erlotinib) (7,8).

Although the therapeutic role of angiogenesis target therapy has been approved in cancer treatment, the way to optimize the dose of angiogenesis inhibitors remains to be determined because of the lack of reliable surrogate markers of tumor angiogenesis. Shaked et al. reported that the levels of circulating endothelial progenitor cells (EPC), which contribute to the tumor vessel formation, reflect the anti-tumor efficacy of anti-angiogenesis regimens (9,10). Growing evidence suggests that the levels of circulating EPC reflect the response to chemotherapy both in animal model and clinical trial (11-13). Thus, circulating EPC can be used as a marker for optimizing and monitoring the anti-angiogenesis therapy including angiogenesis inhibitors and chemotherapy.

Circulating endothelial cells (CEC), especially apoptotic CEC, were observed to increase in breast cancer patients with a clinical benefit (defined as a clinical response or a stable disease) after metronomic therapy (14). Preclinical models indicated that the source of apoptotic CEC was most likely the tumor vasculature (14).

Whether circulating EPC or CEC can be served as markers of CCRT efficacy and toxicity in cervical cancer or not remains undetermined. Since CCRT is now a standard treatment of locally advanced and high-risk cervical cancer, the development of the surrogate marker for monitoring CCRT response and optimize treatment intensity, again, is very important.

ELIGIBILITY:
Inclusion Criteria:

* Receiving chemoradiation

Exclusion Criteria:

* Stage IVB

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cervical cancer stage Ib - IVA
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2007-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Jen Chen, MD,PhD, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan